CLINICAL TRIAL: NCT05109000
Title: Clinical Effects of the Subcutaneous Injection of 10ml of Normal Saline and Bacteriostatic Saline: A Double-Blind Randomized Clinical Trial
Brief Title: Comparison of Subcutaneous Injection of Normal Saline and Bacteriostatic Saline
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jeffrey Alan Klein, MD (Industry)
Responsible Party: Sponsor-Investigator, Jeffrey Alan Klein, MD, Founder and CEO, Physician, HK Surgical, Inc.
Organization: HK Surgical, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NS vs. BS
Record Dates: First submitted 2021-10-13; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Injection Site Irritation; Injection Site Bruising; Injection Site Discomfort; Benzoic Acid Adverse Reaction; Anesthesia, Local
Keywords: normal saline; bacteriostatic saline; subcutaneous injection
MeSH Terms: interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: Subjects will receive both treatments: one in each thigh. Random allocation of subcutaneous injections of 10 mL of normal saline into one anterior thigh and 10 mL of bacteriostatic saline into the contralateral anterior thigh. Paired t-tests to compare the clinical effects of the two solutions.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal Saline (Experimental): This is a randomized, double-blind, single-center clinical trial comparing normal saline and bacteriostatic saline subcutaneous injection within a single subject. In this arm, the subject will receive a 10 mL subcutaneous injection of normal saline into either their left or right anterior thigh. The side will be determined by randomization protocol.
  Interventions: Drug: Sodium Chloride 0.9% Inj
- Bacteriostatic Saline (Experimental): This is a randomized, double-blind, single-center clinical trial comparing normal saline and bacteriostatic saline subcutaneous injection within a single subject. In this arm, the subject will receive a 10 mL subcutaneous injection of bacteriostatic saline into either their left or right anterior thigh. The side will be determined by randomization protocol.
  Interventions: Drug: Bacteriostatic Sodium Chloride 0.9 % INJECTION VIAL (ML)

INTERVENTIONS:
Drug: Sodium Chloride 0.9% Inj — 10 mL subcutaneous injection into one randomized anterior thigh of subject
  Other Names: normal saline
  Arms: Normal Saline
Drug: Bacteriostatic Sodium Chloride 0.9 % INJECTION VIAL (ML) — 10 mL subcutaneous injection into the contralateral anterior thigh of subject
  Other Names: bacteriostatic saline
  Arms: Bacteriostatic Saline

SUMMARY:
This is a randomized, double-blind, single-center clinical trial comparing normal saline and bacteriostatic saline subcutaneous injection within a single subject. While both normal saline and bacteriostatic saline can be administered intravenously, this study aims to investigate their effects following subcutaneous injection. While benzyl alcohol (the bacteriostatic component of bacteriostatic saline) is known to have local anesthetic properties, it also is an irritant and can cause inflammation at the injection site. Based on clinical experience investigators anticipate that a normal saline injection will cause a mild stinging sensation and no subsequent inflammation. In contrast, subcutaneous injection of bacteriostatic saline will not cause stinging but will cause a mild degree of inflammation which is manifested as mild tenderness and mild ecchymosis at the site of injection.

DETAILED DESCRIPTION:
Both normal saline and bacteriostatic saline are often used as vehicles for the injection of therapeutic drugs. However, their properties differ slightly as a result of the 0.9% benzyl alcohol component of BS. While benzyl alcohol is known to have local anesthetic properties, it also is an irritant and can cause inflammation at the injection site. In acidic conditions, benzyl alcohol is converted to benzoic acid and benzaldehyde. Objective and prospective data are needed to confirm these characteristics.

The present protocol calls for random allocation of subcutaneous injections of 10 mL of NS into one anterior thigh and 10 mL of BS into the contralateral anterior thigh. Based on the verified safety of up to 30 mL of 0.9% bacteriostatic saline, this volume of saline solution poses little to no risk.

Each thigh will receive one subcutaneous injection of either NS or BS, which will be determined by random allocation. Clinical follow-up examination will be done at 24 hours, 48 hours, and 7 days.

It is expected that by day seven, all signs of inflammation or bruising will have resolved.

Both NS and BS are FDA-approved for subcutaneous injection and are commonly utilized daily by many physicians. A study documenting the benefits and disadvantages of NS and BS has never been done to the investigators' knowledge and will be helpful for medical professionals in determining which type of solution to use in certain circumstances.

The sample size for this study is 32 subjects with a stopping point for analysis after 16 subjects. The sample size must be a multiple of four to satisfy the randomization in groups of four criteria. Investigators are analyzing the t-statistics at a level of alpha = 0.01, considering the Bonferroni correction. If after 16 subjects, statistical significance showing a difference between NS and BS has not been reached, investigators will continue with 16 more subjects.

Tenderness, soreness, and pruritis NPS will be evaluated by paired t-tests to determine if the effects of injection by NS vs. BS differ at each of the four evaluation times. Investigators will do the same for the quantitative data gathered for bruising and redness surface area. This quantitative analysis will result in t-statistics and corresponding P-values which will be evaluated with an alpha = 0.01, considering the Bonferroni correction. For the categorical data for the intensity of bruising and redness/inflammation, investigators will create the categories of none (0), mild (1), moderate (2), and intense (3) and use this data to perform t-tests for significance.

ELIGIBILITY:
Inclusion Criteria:

1. All volunteer subjects will be healthy, mature in behavior and temperament, and without mental impairment.
2. A volunteer must have signed an informed consent form prior to participation.
3. A subject must be at least 16 years of age.
4. All subjects must weigh at least 40kg = 88lb.
5. All subjects must complete a standard medical history questionnaire.
6. All subjects must agree to return for a follow-up examination, 1 day, 2 days, and 1-week post-injections.

Exclusion Criteria:

* Pregnant women are excluded.
* History of an adverse reaction to percutaneous injections, such as fainting and lightheadedness (vasovagal reactions, near syncope).
* Significant needle phobia or anxiety.
* Vasovagal reaction associated with any medical procedures or the sight of blood.
* History of having or having had a blood-born infection with HIV, Hepatitis B, Hepatitis C.
* Evidence of active skin infection.
* Pre-existing or concurrent Infections (cutaneous, urinary, pneumonia are exclusionary).
* History of radiation therapy or surgery involving the area near the proposed injection site.
* Uncontrolled or labile hypertension.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Injection Pain | Time Post-Injection: 0 minutes
  Numerical Pain Score (NPS): 0-10
Erythema | Time Post-Injection: 5 minutes
  Intensity by visual objective assessment: none (0), mild (1), moderate (2), intense (3)
Erythema | Time Post-Injection: 1 hour
  Intensity by visual objective assessment: none (0), mild (1), moderate (2), intense (3)
Erythema | Time Post-Injection: 24 hours
  Intensity by visual objective assessment: none (0), mild (1), moderate (2), intense (3)
Erythema | Time Post-Injection: 48 hours
  Intensity by visual objective assessment: none (0), mild (1), moderate (2), intense (3)
Erythema | Time Post-Injection: 7 days
  Intensity by visual objective assessment: none (0), mild (1), moderate (2), intense (3)
Bruising | Time Post-Injection: 5 minutes
  Intensity by visual objective assessment: none (0), mild (1), moderate (2), intense (3)
Bruising | Time Post-Injection: 1 hour
  Intensity by visual objective assessment: none (0), mild (1), moderate (2), intense (3)
Bruising | Time Post-Injection: 24 hours
  Intensity by visual objective assessment: none (0), mild (1), moderate (2), intense (3)
Bruising | Time Post-Injection: 48 hours
  Intensity by visual objective assessment: none (0), mild (1), moderate (2), intense (3)
Bruising | Time Post-Injection: 7 days
  Intensity by visual objective assessment: none (0), mild (1), moderate (2), intense (3)
Tenderness | Time Post-Injection: 5 minutes
  Numerical Pain Score (NPS): 0-10
Tenderness | Time Post-Injection: 1 hour
  Numerical Pain Score (NPS): 0-10
Tenderness | Time Post-Injection: 24 hours
  Numerical Pain Score (NPS): 0-10
Tenderness | Time Post-Injection: 48 hours
  Numerical Pain Score (NPS): 0-10
Tenderness | Time Post-Injection: 7 days
  Numerical Pain Score (NPS): 0-10
Soreness | Time Post-Injection: 5 minutes
  Numerical Pain Score (NPS): 0-10
Soreness | Time Post-Injection: 1 hour
  Numerical Pain Score (NPS): 0-10
Soreness | Time Post-Injection: 24 hours
  Numerical Pain Score (NPS): 0-10
Soreness | Time Post-Injection: 48 hours
  Numerical Pain Score (NPS): 0-10
Soreness | Time Post-Injection: 7 days
  Numerical Pain Score (NPS): 0-10

CONTACTS AND LOCATIONS:
Locations (1):
- HK Dermatology, San Juan Capistrano, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers